CLINICAL TRIAL: NCT04191109
Title: Intensive Rehabilitation Program for Subacute Stroke Patients in an Inpatient Rehabilitation Facility: Describing A Protocol Study
Brief Title: BRAIN-CONNECTS: Intensive Rehabilitation Program for Subacute Stroke Patients in an Inpatient Rehabilitation Facility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Esther Duarte, Head of Physical Medicine and Rehabilitation Department, Parc de Salut Mar
Other Study IDs: 34/C/2017- BRAIN-CONNECTS
Record Dates: First submitted 2019-10-29; First posted 2019-12-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: Stroke; Intensive Rehabilitation; Time; Physiotherapy; Occupational Therapy; Speech language therapy
MeSH Terms: conditions — Stroke; Communication Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subacute stroke patients admitted to an inpatient rehabilitation facility.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study in which the amount of therapy performed during the rehabilitation program will be registered.Data regarding feasibility and safety of the program will be also recorded. Indeed, functional, cognitive and quality of life outcomes will be assessed.

SUMMARY:
This is an observational study aiming to describe an intensive rehabilitation program for stroke patients in an inpatient rehabilitation facility, measuring the time and reporting activities performed during the therapy sessions (physiotherapy, occupational and speech language therapy). Indeed, functional and cognitive outcomes will be reported, and data about feasibility and safety of the rehabilitation program will also be recorded.

DETAILED DESCRIPTION:
This is an observational descriptive study that will be performed in an inpatient intensive rehabilitation unit. Stroke patients admitted in our neuro-rehabilitation unit who follow the inclusion criteria, will be invited to participate. The main objective of the study is to register the time spent in different activities during therapy session performed in the intensive rehabilitation program. At the end of each session a sum of the minutes spent in each activity will be performed and at the end of the rehabilitation program the average of time spent in each therapy will be calculated. Indeed, throughout these data the total amount of time spent on rehabilitation (hours and minutes) will be obtained. Secondary objectives are to report changes on functional, cognitive and health status outcomes during different time-frames. This outcomes will be assessed at baseline (admission on neuro-rehabilitation unit), at discharge of rehabilitation unit (average of 30 days after stroke), at 3 months and 6 months after stroke. Safety and Feasibility of the program will also de recorded. Feasibility will be assessed by adherence to the prescribed program, including the register of the following parameters: attendance rate (number of planned sessions attended), training session modification (dose reduction or early termination of the individual session) and reasons for training interruption (2 or more days without training session) as fatigue, dizziness, fever… Safety will be assessed registering any adverse event related to rehab (ie. episodes of falls,..)

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 or over,
2. first-ever intracerebral ischemic or hemorrhagic stroke confirmed by neuroimaging,
3. less than 3 weeks of stroke onset,
4. moderate-to severe impairment (National Institute of Health Stroke Scale [NIHSS] score between 5 and 13),
5. functionally independent prior to stroke (Rankin > 2),
6. no major cognitive deficits affecting comprehension (Mini-Mental State Examination >24), (7) ability to understand Spanish and/or Catalan

Exclusion Criteria:

* Patients with any other neurological or psychiatric condition will be excluded.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subacute stroke patients involved in an inpatient intensive rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-25 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Body Structure and Function: The Fugl-Meyer Assessment-upper limb (FMA-UL) will assess arm impairment. (Fugl-Meyer et al., 1975). | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes in the measurement of arm impairment. Performance is rated on a three point ordinal scale from 0 to 2, with a maximum score of 66, a higher score indicates minimal or no impairment.
Body Structure and Function: Western Aphasia Bedside (WAB) is used to assess the language function of adults with stroke. (Risser, AH et al, 1985) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on WAB will be used to measure language skills. WAB will be used to assess the linguistic skills (information content, fluency, auditory comprehension, repetition, naming and word finding, reading, and writing) and main nonlinguistic skills (drawing, block design, calculation, and praxis) of adults with aphasia.
Body Structure and Function:Cognitive impairment will be assessed using the Montreal Cognitive Assessment (MoCA) (Nasreddine ZS. et al 2005) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on MOCA will be used to detect the cognitive impairments. MOCA is a brief cognitive screening with high sensitivity and specificity for detecting middle cognitive impairment.
Body Structure and Function: Anxiety and Depression that will be assessed using the Hospital Anxiety Depression scale (HADS) (Aben I et al., 2002). | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on psychological distress in stroke patients. HADS consists in in 14 items, which can be divided into two subscales of seven items each: the anxiety subscale (HADS-A) and the depression subscale (HADS-D). The respondent rates each item on a 4-point scale ranging from 0 (absence) - 3 (extreme presence). The total score is out of 42 (21 per subscale).
Body Structure and Function: Apathy will be assessed throughout the Apathy Evaluation Scale. (Marin RS et al. 1993) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on apathy in stroke patients. Thuis is a tool that quantifies and characterise apathy in adult patients. The AES, which uses 18 specific items to quantify apathy within a scoring range of 18 to 72.
Body Structure and Function: Limb strength will assessed using the Motricity Index Motricity Index (MI) (Collin C et al.1990). | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on upper and lower limb strength using MI which is an ordinal method of measuring limb strength, this test has 6 items on each side 3 for the arm and 3 for the leg.
Activity Level: Assessment of functional disability in basic activities of daily living will be performed using Barthel Index (BI). (Mahoney FI et al.,1965) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on functional disability of stroke patients using BI, which evaluates 10 basic activities of self-care (feeding, grooming, dressing, toileting, bathing, and continence of bowel and bladder) and mobility (transferring, walking, stair climbing) on a total score from 0 (totally dependent) to 100 (totally independent) functioning.
Activity Level: Disability level will be assessed throughout modified Ranking scale (MRS) (Van Swieten JC et al., 1988, Bonita R et al., 1988) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Change in the disability level after stroke. The MRS is a global outcome rating scale ranging from 0 (no impairment) to 5 (bedridden, incontinent, requiring constant nursing care and attention) and 6 (fatal outcome).
Activity Level: Gait speed on 10m walking test. (Pohl M et al., 2007) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on gait speed will be assessed during a 10 meter walking test
Activity Level: Arm function will assessed using the Action Research Arm Test (ARAT) (Hsieh CL et al., 1998, Lang CE et al., 2006) | Admission on rehabilitation unit - Average 30 days after stroke (discharge of rehabilitation unit) - 3 months and 6 months after stroke
  Changes on arm function will be reported throughout ARAT, this assessment is divided into four sub tests of grasp, grip, pinch and gross arm movement. Performance on each item is rated on a four-point ordinal scale from 0 to 3 with a maximum score of 57, a higher score indicating a better level of function.
Participation Level will be assessed throughout the Stroke Impact Scale (SIS). (Richardson M et al., 2016, Duncan PW et al., 1999) | At 3 months and 6 months after stroke
  Changes on Health related quality of life will be assessed throughout SIS , that is a 59-item measurement, which assess 8 domains (strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking and participation level). Each item is rated in a 5 point likert scale in terms of difficulty the patient has experienced in completing each item. Summative scores are generated for each domain, scores ranges from 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duarte, PhD, Principal Investigator — Parc de Salut Mar - Hospital del Mar i de L´Esperança
Locations (1):
- Parc de Salut Mar - Hospital del Mar i de L´Esperança, Barcelona, Spain

REFERENCES:
- [Derived] Sartor MM, Grau-Sanchez J, Guillen-Sola A, Boza R, Puig J, Stinear C, Morgado-Perez A, Duarte E. Intensive rehabilitation programme for patients with subacute stroke in an inpatient rehabilitation facility: describing a protocol of a prospective cohort study. BMJ Open. 2021 Oct 18;11(10):e046346. doi: 10.1136/bmjopen-2020-046346. PMID 34663650